CLINICAL TRIAL: NCT01159951
Title: Time Trend Analysis of the Incidence of Hepatitis- Related Outcomes (Viral Hepatitis A and Unspecified Viral Hepatitis) Reported to the Surveillance System of Panama, 2000-2010
Brief Title: Analysis of Trends Over Time of Hepatitis Related Incidence in Panama
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112263
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — No samples retained

GROUPS / COHORTS (1):
- Hepatitis Cohort: Subjects suffering with hepatitis
  Interventions: Other: Epidemiologic Surveillance System of the Ministry of Health of Panama

INTERVENTIONS:
Other: Epidemiologic Surveillance System of the Ministry of Health of Panama — Systematic review of the databases of epidemiologic surveillance system, Ministry of health, Panama

SUMMARY:
The purpose of this study is to analyze the incidence of baseline hepatitis related outcomes (viral hepatitis A and unspecified viral hepatitis) together with the current frequency of the same outcome after introduction of Havrix™ in Panama.

DETAILED DESCRIPTION:
In this study, systematic review of the databases of epidemiologic surveillance system (Ministry of Health), for hepatitis related outcomes will be performed. The analysis will be performed by age group, years and country region.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis related outcomes occurred during the period analyzed and registered in the Epidemiologic Surveillance System of the Ministry of Health, will be collected for the study

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population to be studied will be all subjects reported with hepatitis related outcomes to the Epidemiologic Surveillance System of the Ministry of Health of Panama, between 2000 and 2010.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of reported hepatitis related outcomes (viral hepatitis A and unspecified viral hepatitis) | In post vaccine introduction period (2008-2010) compared to pre-vaccination period (2000-2007)

SECONDARY OUTCOMES:
Occurrence of hepatitis related outcomes (viral hepatitis A and unspecified viral hepatitis) by year | From year 2000 until year 2010
Occurrence of hepatitis related outcomes (viral hepatitis A and unspecified viral hepatitis) by age groups | From year 2000 until year 2010
Occurrence of hepatitis related outcomes (viral hepatitis A and unspecified viral hepatitis) by region | From year 2000 until year 2010

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Clayton, Provincia de Panamá, Panama

REFERENCES:
- [Derived] Estripeaut D, Contreras R, Tinajeros O, Castrejon MM, Shafi F, Ortega-Barria E, DeAntonio R. Impact of Hepatitis A vaccination with a two-dose schedule in Panama: Results of epidemiological surveillance and time trend analysis. Vaccine. 2015 Jun 22;33(28):3200-7. doi: 10.1016/j.vaccine.2015.04.100. Epub 2015 May 14. PMID 25981490